CLINICAL TRIAL: NCT04615923
Title: HEALEY ALS Platform Trial - Regimen D Pridopidine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merit E. Cudkowicz, MD (Other)
Collaborators: Prilenia (Industry)
Responsible Party: Sponsor-Investigator, Merit E. Cudkowicz, MD, Chief, Neurology Department, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P003518D
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Results first posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Placebo-Controlled; Double-Blind; Regimen Specific Appendix; Lou Gehrig's Disease; Pridopidine; Prilenia Therapeutics
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — pridopidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pridopidine (Experimental): Pridopidine is administered orally twice daily for 24 weeks.
  Interventions: Drug: Pridopidine
- Matching Placebo (Placebo Comparator): Matching placebo is administered orally twice daily for 24 weeks.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Pridopidine — Administration: Oral
  Dose: 45mg twice daily
  Arms: Pridopidine
Drug: Matching Placebo — Administration: Oral
  Dose: one capsule twice daily
  Arms: Matching Placebo

SUMMARY:
The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS.

Regimen D will evaluate the safety and efficacy of a single study drug, pridopidine, in participants with ALS.

DETAILED DESCRIPTION:
The HEALEY ALS Platform Trial is a perpetual multi-center, multi-regimen clinical trial evaluating the safety and efficacy of investigational products for the treatment of ALS. This trial is designed as a perpetual platform trial. This means that there is a single Master Protocol dictating the conduct of the trial. The HEALEY ALS Platform Trial Master Protocol is registered as NCT04297683.

Once a participant enrolls into the Master Protocol and meets all eligibility criteria, the participant will be eligible to be randomized into any currently enrolling regimen. All participants will have an equal chance of being randomized to any currently enrolling regimen.

If a participant is randomized to Regimen D Pridopidine, the participant will complete a screening visit to assess additional Regimen D eligibility criteria. Once Regimen D eligibility criteria are confirmed, participants will complete a baseline assessment and be randomized in a 3:1 ratio to either active pridopidine or matching placebo.

Regimen D will enroll by invitation, as participants may not choose to enroll in Regimen D. Participants must first enroll into the Master Protocol and be eligible to participate in the Master Protocol before being able to be randomly assigned to Regimen D.

For a list of enrolling sites, please see the HEALEY ALS Platform Trial Master Protocol under NCT04297683.

ELIGIBILITY:
Inclusion Criteria:

* No additional inclusion criteria beyond the inclusion criteria specified in the Master Protocol (NCT NCT04297683).

Exclusion Criteria:

* The following exclusion criteria are in addition to the exclusion criteria specified in the Master Protocol (NCT NCT04297683).

  1. Participants with a confirmed prolonged Fridericia-corrected QT (QTcF) interval (defined as a QTcF interval of >450 ms for men and >470 ms for women).
  2. Participants with clinically significant heart disease, clinically significant history of arrhythmia, symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia, or presence of left bundle branch block.
  3. Participants with known history of long QT syndrome or a first degree relative with this condition.
  4. Participants using prohibited medications within the 4 weeks prior to the Regimen Specific Screening Visit, as detailed in section 5.9.
  5. Participants using the following medications at the time of the Regimen Specific Screening Visit:

     1. Nuedexta - at a dosage higher than 20 mg dextromethorphan + 10 mg quinidine BID
     2. Citalopram - at a dosage higher than 20 mg/day
     3. Escitalopram - at a dosage higher than 10 mg/day
  6. Participants with a known allergy to any ingredient of the study intervention (pridopidine, silicified microcrystalline cellulose, and magnesium stearate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Healey Center for ALS at Mass General, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Writing Committee for the HEALEY ALS Platform Trial; Shefner JM, Oskarsson B, Macklin EA, Chibnik LB, Quintana M, Saville BR, Detry MA, Vestrucci M, Marion J, McGlothlin A, Heiman-Patterson T, Chase M, Pothier L, Harkey BA, Yu H, Sherman AV, Hall M, Kittle G, Berry JD, Babu S, Andrews J, D'Agostino D, Tustison E, Scirocco E, Giacomelli E, Alameda G, Locatelli E, Ho D, Quick A, Ajroud-Driss S, Katz J, Heitzman D, Appel SH, Shroff S, Felice K, Maragakis NJ, Simmons Z, Miller TM, Olney N, Weiss MD, Goutman SA, Fernandes JA, Jawdat O, Owegi MA, Foster LA, Vu T, Ilieva H, Newman DS, Arcila-Londono X, Jackson CE, Ladha S, Caress JB, Swenson A, Peltier A, Lewis RA, Fee D, Elliott M, Bedlack R, Kasarskis EJ, Elman L, Rosenfeld J, Walk D, McIlduff C, Twydell P, Young E, Johnson K, Rezania K, Goyal NA, Cohen JA, Benatar M, Jones V, Shah J, Beydoun SR, Wymer JP, Zilliox L, Nayar S, Pattee GL, Martinez-Thompson J, Leitner ML, Chen K, Goldberg YP, Cohen Y, Geva M, Hayden MR, Paganoni S, Cudkowicz ME; HEALEY ALS Platform Trial Study Group. Pridopidine in Amyotrophic Lateral Sclerosis: The HEALEY ALS Platform Trial. JAMA. 2025 Feb 17;333(13):1128-37. doi: 10.1001/jama.2024.26429. Online ahead of print. PMID 40067755

RESULTS

PARTICIPANT FLOW:
Groups:
- Pridopidine: Pridopidine is administered orally twice daily for 24 weeks.
  Pridopidine: Administration: Oral
  Dose: 45mg twice daily
- Matching Placebo: Matching placebo is administered orally twice daily for 24 weeks.
  Matching Placebo: Administration: Oral
  Dose: one capsule twice daily
Period: Overall Study
Arm/Group | Pridopidine | Matching Placebo
Started | 120 | 42
Completed | 96 | 38
Not Completed | 24 | 4

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes only placebo participants from the Regimen D Efficacy Regimen Only (ERO) sample; shared placebo participants from other regimens are not included in the Baseline Analysis Population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pridopidine | Matching Placebo | Total
Number analyzed (Participants) | 120 | 42 | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (10.10) | 57.1 (9.86) | 57.7 (10.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 9 | 57
  Male | 72 | 33 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 1 | 12
  Not Hispanic or Latino | 107 | 41 | 148
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 105 | 39 | 144
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 2
El Escorial Diagnosis [Count of Participants; unit: Participants]
  Clinically Definite ALS | 50 | 18 | 68
  Clinically Probable ALS | 40 | 12 | 52
  Clinically Probable ALS - Laboratory Supported | 22 | 5 | 27
  Clinically Possible ALS | 8 | 7 | 15
ALS Onset Location [Count of Participants; unit: Participants]
  Axial | 1 | 2 | 3
  Bulbar | 23 | 10 | 33
  Generalized | 2 | 0 | 2
  Limb | 93 | 30 | 123
  Multiple | 1 | 0 | 1
Baseline Edaravone Use Flag [Count of Participants; unit: Participants]
  No | 92 | 32 | 124
  Yes | 28 | 10 | 38
Baseline Riluzole Use Flag [Count of Participants; unit: Participants]
  No | 30 | 9 | 39
  Yes | 90 | 33 | 123
Kings Stage [Count of Participants; unit: Participants] — The King's ALS Clinical Staging System is a 4-level ordinal scale with the first three levels indicating the number (1, 2, or 3) of distinct central nervous system regions (bulbar, upper limb, and lower limb) with neuromuscular dysfunction. Level 4a indicates nutritional failure and level 4b indicates respiratory failure. Higher scores indicate a worse disease state.
  Participants
    1 Region with Neuromuscular Dysfunction | 21 | 7 | 28
    2 Regions with Neuromuscular Dysfunction | 36 | 7 | 43
    3 Regions with Neuromuscular Dysfunction | 31 | 18 | 49
    4a/4b Nutritional/Respiratory Failure | 32 | 10 | 42
ALSFRS-R Total Score [Mean (Standard Deviation); unit: points] — The ALS Functional Rating Score-Revised (ALSFRS-R) measures 12 aspects of physical function. Each of the 12 questions assessing distinct functional ability is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function.
  points | 34.3 (6.71) | 35.0 (7.07) | 34.5 (6.79)
Baseline Decline in ALSFRS-R [Mean (Standard Deviation); unit: points per month] — The ALS Functional Rating Score-Revised (ALSFRS-R) measures 12 aspects of physical function. Each of the 12 questions assessing distinct functional ability is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function.
  Baseline is divided by the number of months between onset of weakness due to ALS and the date of Baseline.
  A higher number indicates greater decline.
  points per month | 0.77 (0.5) | 0.71 (0.455) | 0.75 (0.488)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.1 (4.63) | 25.9 (4.07) | 26.1 (4.48)
Delay in ALS Symptom Onset and Diagnosis [Mean (Standard Deviation); unit: months] | 10.5 (6.34) | 10.4 (6.50) | 10.5 (6.36)
SVC [Mean (Standard Deviation); unit: percent predicted] — Population: Number analyzed in row differs from overall number due to missing data.
  percent predicted
    number analyzed (Participants) | 116 | 42 | 158
    (all) | 78.3 (17.35) | 77.5 (16.72) | 78.1 (17.13)
Serum Cereatinine Concentration [Mean (Standard Deviation); unit: mg/dL] | 0.7 (0.19) | 0.8 (0.18) | 0.7 (0.19)
Time Since Symptom Onsent at Baseline (Months since ALS symptom onset) [Mean (Standard Deviation); unit: months] | 20.6 (8.16) | 21.6 (10.0) | 20.8 (8.65)
Weight [Mean (Standard Deviation); unit: kg] | 76.6 (15.92) | 79.3 (15.63) | 77.3 (15.84)
Serum NfL Concentration [Mean (Standard Deviation); unit: ng/L] — Population: Number analyzed in row differs from overall number due to missing data.
  ng/L
    number analyzed (Participants) | 119 | 40 | 159
    (all) | 92.7 (61.24) | 114.6 (73.25) | 98.2 (64.93)

OUTCOME MEASURES:

1. Primary Outcome: Disease Progression as Assessed by the ALSFRS-R Total Score
Description: Change in disease severity over time as measured by the ALS Functional Rating Scale-Revised (ALSFRS-R). Each type of function is scored from 4 (normal) to 0 (no ability), with a maximum total score of 48 and a minimum total score of 0. Patients with higher scores have more physical function.
Time Frame: Baseline to 24 Weeks
Population: Outcome measure data was analyzed using the Full Analysis Set, which included shared placebo from other regimens, as pre-specified in the Regimen Statistical Analysis Plan. Regimen A (NCT04436497), Regimen B (NCT04436510) and Regimen C (NCT04414345) contributed placebo participants into the shared placebo cohort used for analysis.
Measure: Mean (Standard Deviation); unit: points per month
Arm/Group | Pridopidine | Matching Placebo
Number analyzed (Participants) | 120 | 162
points per month | -0.99 (0.077) | -1.00 (0.070)
Statistical Analysis 1: Comparison: Pridopidine vs Matching Placebo; Test type: Superiority; Bayesian shared-parameter model — Posterior probability that the disease rate ratio (DRR) is less than 1 (i.e. Pridopidine slowed progression) was (0.5475). NOTE: p-value is not provided for Bayesian model; A Bayesian shared-parameter model of change in disease severity as measured by ALSFRS-R total score and mortality; Disease Rate Ratio = 0.99, 95% CI 2-sided [0.801 to 1.207], Standard Deviation 0.103 — DDR <1 imply slowing of disease progression by verdiperstat relative to placebo.Note: reported "Confidence Interval" is actually a Bayesian credible interval; The DRR parameter for active treatment represents the relative change to the rate of decline of ALSFRS-R and the rate of mortality of treated participant relative to a placebo participant. The estimated DRR can also be interpreted as the average rate of decline in function and mortality. The model includes covariates for baseline use of edaravone, baseline use of riluzole, months since onset of symptoms, and pre-baseline slope of ALSFRS-R, and random effects for regimen and participant-specific slopes

2. Primary Outcome: Mortality Event Rate
Description: Mortality is defined as death or death equivalent. A participant is determined to meet the criteria of death equivalent if permanent assisted ventilation (PAV) is used for more than 22 hours per day for more than seven days in a row. The rate of mortality was estimated from a Bayesian shared-parametric model that assumed exponentially distributed survival times.
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: events per month
Arm/Group | Pridopidine | Matching Placebo
Number analyzed (Participants) | 120 | 162
events per month | 0.012 (0.0029) | 0.012 (0.0029)

3. Secondary Outcome: Change in Bulbar Function in Participants With Bulbar Dysfunction at Baseline
Description: Change in bulbar function over time in participants with bulbar dysfunction at baseline as measured by the ALS Functional Rating Scale-Revised (ALSFRS-R) bulbar subdomain. Each question is scored from 4 (normal) to 0 (no ability), with a maximum total score of 12 and a minimum total score of 0 for the bulbar subdomain. Patients with higher scores have more bulbar function.
  Participants were classified as having bulbar dysfunction at baseline if their score on the ALSFRS-R bulbar domain (Q1-Q3) score was less than 12.
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: point change from baseline
Arm/Group | Pridopidine | Matching Placebo
Number analyzed (Participants) | 75 | 103
point change from baseline | -1.78 (0.261) | -1.69 (0.210)
Statistical Analysis 1: Comparison: Pridopidine vs Matching Placebo; Test type: Superiority; p = 0.78, Mixed Models Analysis; Covariates include baseline use of edaravone and riluzole, months since symptom onset, and pre-baseline ALSFRS-R slope; Median Difference (Net) = -0.09, 95% CI 2-sided [-0.75 to 0.57], Standard Error of Mean 0.334 — Pridopidine 24-week change from baseline relative to placebo 24-week change from baseline

4. Secondary Outcome: Bulbar Function in All Randomized Participants
Description: Change in bulbar function over time in all randomized participants as measured by the ALS Functional Rating Scale-Revised (ALSFRS-R) bulbar subdomain. Each question is scored from 4 (normal) to 0 (no ability), with a maximum total score of 12 and a minimum total score of 0 for the bulbar subdomain. Patients with higher scores have more bulbar function.
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: point change from baseline
Arm/Group | Pridopidine | Matching Placebo
Number analyzed (Participants) | 120 | 162
point change from baseline | -1.16 (0.169) | -1.25 (0.141)
Statistical Analysis 1: Comparison: Pridopidine vs Matching Placebo; Test type: Superiority; p = 0.6594, Mixed Models Analysis; Covariates include baseline use of edaravone and riluzole, months since symptom onset, and pre-baseline ALSFRS-R slope; Median Difference (Net) = 0.10, 95% CI 2-sided [-0.33 to 0.52], Standard Error of Mean 0.217 — Pridopidine 24-week change from baseline relative to placebo 24-week change from baseline

5. Secondary Outcome: Respiratory Function
Description: Change in respiratory function over time as measured by Slow Vital Capacity (SVC).
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Pridopidine | Matching Placebo
Number analyzed (Participants) | 120 | 162
percent change | -8.81 (1.351) | -8.35 (1.132)
Statistical Analysis 1: Comparison: Pridopidine vs Matching Placebo; Test type: Superiority; p = 0.7918, Mixed Models Analysis; Covariates include baseline use of edaravone and riluzole, months since symptom onset, and pre-baseline ALSFRS-R slope; Mean Difference (Net) = -0.46, 95% CI 2-sided [-3.89 to 2.96], Standard Error of Mean 1.745 — Pridopidine 24-week change from baseline relative to placebo 24-week change from baseline

6. Secondary Outcome: Bulbar Function in Participants With Rapid Pre-baseline Progression
Description: Change in bulbar function over time in participants with rapid pre-baseline progression as measured by the ALS Functional Rating Scale-Revised (ALSFRS-R) bulbar subdomain. Each question is scored from 4 (normal) to 0 (no ability), with a maximum total score of 12 and a minimum total score of 0 for the bulbar subdomain. Patients with higher scores have more bulbar function.
  Participants were classified with rapid pre-baseline progression if their change in ALSFRS-R total score between Master Protocol Screening and Regimen Baseline was greater than or equal or 0.75 points per month.
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: points change from baseline
Arm/Group | Pridopidine | Matching Placebo
Number analyzed (Participants) | 51 | 48
points change from baseline | -1.54 (0.297) | -1.54 (0.302)
Statistical Analysis 1: Comparison: Pridopidine vs Matching Placebo; Test type: Superiority; p = 0.9903, Mixed Models Analysis; Covariates include baseline use of edaravone and riluzole, months since symptom onset, and pre-baseline ALSFRS-R slope; Median Difference (Net) = 0.01, 95% CI 2-sided [-0.83 to 0.84], Standard Error of Mean 0.426 — Pridopidine 24-week change from baseline relative to placebo 24-week change from baseline

7. Secondary Outcome: Time to Bulbar Decline
Description: Time to first decline of 1-point or greater post baseline in the ALSFRS-R bulbar domain score among all participants.
  Analysis performed using interval-censored survival analysis. Results presented as median interval (upper & lower bounded) time to event.
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pridopidine | Matching Placebo
Number analyzed (Participants) | 120 | 162
days
  Lower Bound of Interval | 84 [53 to 141] | 66 [56 to 105]
  Upper Bound of Interval | 86 [83 to 141] | 77 [68 to 115]
Statistical Analysis 1: Comparison: Pridopidine vs Matching Placebo; Test type: Superiority — Analysis performed using interval-censored survival analysis. This type of model accommodates interval censoring between ALSFRS-R assessments; Regression, Cox; Interval censored cox model adjusted for time since symptom onset, pre-baseline change in ALSFRS-R, baseline use of edaravone, riluzole, and neudexta; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.69 to 1.27]

8. Secondary Outcome: Muscle Strength
Description: Change in muscle strength over time as measured isometrically using hand-held dynamometry (HHD).
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Pridopidine | Matching Placebo
Number analyzed (Participants) | 120 | 162
percent change | -26.74 (2.556) | -24.97 (2.123)
Statistical Analysis 1: Comparison: Pridopidine vs Matching Placebo; Test type: Superiority; p = 0.5888, Mixed Models Analysis; Covariates include baseline use of edaravone and riluzole, months since symptom onset, and pre-baseline ALSFRS-R slope; Mean Difference (Net) = -1.78, 95% CI 2-sided [-8.23 to 4.67], Standard Error of Mean 3.285 — Pridopidine 24-week change from baseline relative to placebo 24-week change from baseline

9. Secondary Outcome: Number of Participants That Experienced Death or Death Equivalent
Description: The number of participants who died or met the criterion for a death equivalent from the date of their baseline visit to the end of the Week 24visit window (generally 175 days after baseline). The death equivalent criterion is use of permanent assisted ventilation (PAV) for more than 22 hours per day for more than 7 days in a row.
Time Frame: Baseline to 24 Weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Pridopidine | Matching Placebo
Number analyzed (Participants) | 120 | 162
Participants | 5 | 6
Statistical Analysis 1: Comparison: Pridopidine vs Matching Placebo; Test type: Superiority; p = 0.9690, Log Rank

ADVERSE EVENTS:
Time Frame: Up to 35 weeks after participant signed Master Protocol consent.
Description: The total at risk number for serious adverse events and other adverse events differs from the overall numbers due to a participant excluded from full analysis set for efficacy analyses and baseline characteristics due to a diagnosis other than ALS in one participant and due to participant included in the full analysis set for efficacy analyses and baseline characteristics due to being randomized but who never initiated study drug and thus was not considered as risk for safety outcomes.
Arm/Group | Pridopidine | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 2/120 | 0/42
Serious Adverse Events (participants affected / at risk) | 16/121 | 3/41
Other Adverse Events (participants affected / at risk) | 106/121 | 37/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pridopidine (N=121) | Matching Placebo (N=41)
Amyotrophic lateral sclerosis (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pridopidine (N=121) | Matching Placebo (N=41)
Muscular weakness (Nervous system disorders) | 29 (33) | 13 (21)
Neuromyopathy (Nervous system disorders) | 24 (37) | 3 (3)
Dysarthria (Nervous system disorders) | 10 (10) | 4 (5)
Dizziness (Nervous system disorders) | 9 (10) | 4 (5)
Headache (Nervous system disorders) | 6 (7) | 1 (1)
Muscle contractions involuntary (Nervous system disorders) | 4 (4) | 3 (4)
Cognitive disorder (Nervous system disorders) | 3 (3) | 3 (3)
Constipation (Gastrointestinal disorders) | 14 (18) | 8 (9)
Diarrhoea (Gastrointestinal disorders) | 15 (22) | 4 (5)
Nausea (Gastrointestinal disorders) | 15 (18) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 13 (13) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 10 (10) | 3 (3)
Salivary hypersecretion (Gastrointestinal disorders) | 10 (10) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 34 (65) | 12 (28)
Contusion (Injury, poisoning and procedural complications) | 8 (11) | 3 (6)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (2) | 4 (6)
Fatigue (General disorders) | 12 (14) | 5 (5)
Oedema peripheral (General disorders) | 9 (10) | 3 (4)
Complication associated with device (General disorders) | 7 (8) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
COVID-19 (Infections and infestations) | 12 (12) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (12) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (13) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Anxiety (Psychiatric disorders) | 8 (8) | 4 (4)
Insomnia (Psychiatric disorders) | 9 (10) | 1 (1)
Depression (Psychiatric disorders) | 6 (6) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/23/NCT04615923/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT04615923/SAP_001.pdf